CLINICAL TRIAL: NCT07304934
Title: A Single-arm, Prospective, Multi-center Cohort Study Based on Deep Learning-based cfDNA Fragment Omics to Verify the TuFEst Model for the Staging Diagnosis of Breast Cancer Lesions and Lymph Nodes
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1028
Record Dates: First submitted 2025-11-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; cfDNA; TuFEst model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Detect tumor-related cfDNA fragments in plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Breast cancer patients who have undergone radical surgery and have not received neoadjuvant therapy
  Interventions: Other: No Intervention: Observational Cohort
- 2: Patients with newly diagnosed invasive breast cancer and confirmed axillary lymph node metastasis, who are willing to undergo radical surgery after treatment (Exploratory Analysis Cohort)
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
Through the research of this project, we expect to achieve the cfDNA fragment omics liquid biopsy technology based on deep learning, verify the accuracy of the TuFEst model in predicting the tumor burden status of breast cancer lesions and lymph nodes in newly diagnosed breast cancer patients and those receiving neoadjuvant therapy, and provide a theoretical basis for large-scale clinical application in the future

DETAILED DESCRIPTION:
1. Based on the previously established TuFEst model, the cfDNA fragment omics liquid biopsy technology based on deep learning is utilized to predict the tumor burden status of breast cancer lesions and lymph nodes, thereby enhancing the accuracy of early diagnosis of breast cancer: This study will collect and analyze blood samples from breast cancer patients at different stages, and use deep learning-based cfDNA fragment omics liquid biopsy technology to extract tumor-related cfDNA fragments and construct a cfDNA fragment omics feature library. Predictions are made based on the TuFEst model. Then, accuracy matching and evaluation are carried out according to the prediction results and the actual breast cancer lesion and lymph node tumor burden status. Verify the efficacy of the TuFEst model in the staging diagnosis of breast cancer.
2. To evaluate the sensitivity, specificity, accuracy and repeatability of the TuFEst model to determine its reliability in clinical application: This study will collect a larger number of blood samples from breast cancer patients based on the previous retrospective cohort to assess the performance of the model in a larger sample prospective cohort. This study will also explore the application of this technology in the monitoring of neoadjuvant therapy for breast cancer, specifically evaluating its application in post-treatment staging diagnosis of breast cancer, prediction of treatment effects, and monitoring of tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70;
2. Direct Surgery Group (Cohort 1) : Radical surgery was performed without neoadjuvant therapy;
3. Neoadjuvant therapy group (Cohort 2) : The initial diagnosis was invasive breast cancer with confirmed axillary lymph node metastasis, and the patient was willing to undergo radical surgery at the end of treatment;
4. Plasma from patients during treatment can be obtained;
5. Be willing to sign the informed consent form. -

Exclusion Criteria:

1. Be pregnant or breastfeeding;
2. Patients whose lesions have been resected;
3. Suffered from other types of malignant tumors with a clear pathological diagnosis within 5 years prior to enrollment;
4. Within the past year of enrollment, the patient had other malignant tumors suspected by imaging, but they were not confirmed by pathology;
5. Suspected distant metastatic lesions on imaging, or potential lymph node lesions that cannot be completely cured by surgery;
6. Have received any blood product infusion treatment in the past 30 days. -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who have been treated at the Second Affiliated Hospital of Zhejiang University School of Medicine (Other Centers) from the date of ethical approval until December 31, 2027
Sampling Method: Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of the TuFEst-based classifier for predicting pathologic node-negative status (pN0) | up to 2 weeks
  Validate the accuracy of the TuFEst model in predicting breast cancer lesion and lymph node tumor burden status among patients with primary breast cancer and those undergoing neoadjuvant therapy.

IPD SHARING:
Plan to Share IPD: No